CLINICAL TRIAL: NCT03158142
Title: The Influence of Atropine on Choroidal Thickness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York College of Optometry (Other)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1000533-1
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atropine group (Experimental): One drop of Atropine Sulfate 1% Oph Soln will be administered either in the morning or at night in each eye. Study measurements will be taken approximately after 1, 12, 24 and 96 hours after drop instillation. After a 2 week wash out period with no eye drops, another drop of 1% atropine sulfate ophthalmic eye drops will be administered either in the morning or night (the visit that was not taken before) and study measurements will be scheduled approximately after 1, 12 24 and 96 hours after drop instillation
  Interventions: Drug: Atropine Sulfate 1% Oph Soln

INTERVENTIONS:
Drug: Atropine Sulfate 1% Oph Soln — Atropine sulphate 1% ophthalmic solution is both a mydriatic and cycloplegic
  Other Names: 1% atropine eye drops

SUMMARY:
Atropine eye drops are increasingly prescribed for the management of progressive myopia or short-sightedness. A previous study suggested that the back of the eye or choroid may be a part of the mechanism by which it induces its effects.

The aim of this study is to characterize the effects of atropine on choroidal thickness and the influence of time of administration (am vs pm). It is hypothesized that the atropine's effect on choroidal thickness will vary with baseline thickness related to diurnal rhythm, where thicker baseline thickness will show a reduced choroidal response.

DETAILED DESCRIPTION:
Atropine eye drops are increasingly prescribed for the management of progressive myopia or short-sightedness. A previous study suggested that the back of the eye or choroid may be a part of the mechanism by which it induces its effects. The choroid shows diurnal variation and the efficacy of atropine on myopia control in relationship to the patient's baseline choroidal thickness is unknown. Thus, the objective of this study is to provide data to characterize the influence of atropine on choroid thickness. The study aims are to:

1. Determine the effect of am or pm atropine application on choroid thickness
2. Determine the effect of atropine on choroid thickness in relationship to baseline thickness

Participants will be asked to attend a screening session and 13 study visits. Following the screening visit, participants will be scheduled to return for 4 visits across 12 hours (4 hour intervals starting from 8am) in a single day where eye shape measurements will be taken to characterize diurnal variations in eye shape.

Subjects will then be randomized to receive a drop of 1% atropine eye drops in both eyes in the morning or a night. Measurements of the shape of the front and back of the eye will be taken after approximately 1, 12, 24 and 96 hours after drop instillation. After a 2 week washout period, 1% atropine eye drops will be administered either in the morning or at night (the visit that was not previously scheduled) and measurements of the shape of the front and back of the eye will be taken after approximately 1, 12, 24 and 96 hours after drop instillation.

ELIGIBILITY:
Inclusion Criteria:

* Good general and ocular health
* Soft contact lens wearers to cease lens wear for at least 24 hours
* No previous rigid gas permeable lens wear

Exclusion Criteria:

* History of ocular surgery, including refractive surgery
* Amblyopia
* Use of ocular medications
* Known allergies or sensitivity to atropine
* Pregnant, plan to become pregnant, or are breastfeeding
* Taking monoamine oxidase inhibitors (MAOIs)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Choroidal thickness | Baseline, then after approximately 1, 12, 24 and 96 hours after atropine instillation
  Change in choroidal thickness after atropine

CONTACTS AND LOCATIONS:
Locations (1):
- State University of New York College of Optometry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
All IPD collected from the study will be made available to other the investigators that have been listed on this study. IPD will be de-identified before making it available to the other investigators. IPD will become available after the end of study data collection. Deidentified IPD will be obtained by other investigator in excel files sent by the primary investigator